CLINICAL TRIAL: NCT05518097
Title: Effects of Central Sensitization on Response to Conventional Physical Therapy in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Haydar Gok, Professor Doctor, Ankara University
Other Study IDs: 10-795-19
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; Neuropathic pain; Central sensitization; Physical therapy; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Neuralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conventional Physical Therapy Program: Patients with knee osteoarthritis underwent a conventional physical therapy program including hotpack, US, TENS and exercise.
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Conventional physical therapy program — Patients with knee osteoarthritis underwent a total of 15 sessions of conventional physical therapy program including hotpack, US, TENS, and exercise 5 days a week, for 3 weeks. Hot pack was applied for 10 minutes, ultrasound was applied continuously at 1 MHz, 1.0 W/cm2 for 10 minutes, and TENS was applied for 30 minutes according to the patient's tolerance. The exercise program consisted of an active, active-assisted range of motion and isometric quadriceps strength training.

SUMMARY:
The aim of this study was to investigate the relationship between central sensitization (CS) and poor response to conventional physical therapy in patients with knee osteoarthritis (OA) by evaluating clinical parameters of pain and functionality.

84 knee OA patients with knee pain for at least 3 months and 30 healthy controls were included in the study. Socio-demographic features of the participants such as age, sex, body mass index (BMI), and duration of symptoms were recorded. Structural damage was assessed by knee radiography. Knee pain and functional status were evaluated by visual analogue scale (VAS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at baseline and immediately after the treatment. Additionally, the following measures were applied at baseline: Central Sensitization Inventory (CSI), Beck Depression Inventory (BDI), Insomnia Severity Index (ISI), Pain Catastrophization Scale (PCS), and PainDETECT Questionnaire (PD-Q). Pressure pain threshold (PPT) was measured with a digital algometer at the painful joint, near the joint area, and in a painless remote region. Patients with knee OA underwent a total of 15 sessions of conventional physical therapy program including hotpack, ultrasound (US), transcutaneous electrical nerve stimulation (TENS), and exercise 5 days a week, for 3 weeks. The control group had no treatment except for the PPT measurement to obtain the reference PPT values. After the treatment, the patients were divided into two groups as 'responders' and 'non-responders' according to their response to treatment. The relationship between the response to physical therapy and clinical parameters was evaluated.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the relationship between central sensitization (CS) and poor response to conventional physical therapy in patients with knee osteoarthritis (OA) by evaluating clinical parameters of pain and functionality.

The study was planned as a prospective, cohort study. Patients presenting with knee pain lasting more than 3 months and diagnosed with primary knee OA according to the American College of Rheumatology (ACR) criteria were screened to be included in the study at the Department of Physical Medicine and Rehabilitation, Ankara University, Faculty of Medicine. The protocol was approved by the Ankara University Faculty of Medicine Clinical Research Ethics Committee (27.05.2019 and Decision No. 10-795-19) and the trial was conducted in accordance with the Declaration of Helsinki and the International Conference on Harmonization Good Clinical Practice Guidelines.

Patients in the OA group underwent a total of 15 sessions of conventional physical therapy program including hotpack, ultrasound (US), transcutaneous electrical nerve stimulation (TENS), and exercise 5 days a week, for 3 weeks. Hot pack was applied for 10 minutes, US was applied continuously at 1 megahertz (MHz), 1.0 W/cm2 for 10 minutes, and TENS was applied for 30 minutes according to the patient's tolerance. The exercise program consisted of an active, active-assisted range of motion and isometric quadriceps strength training. The control group had no treatment except for the PPT measurements to obtain the reference PPT values. At the end of treatment, patients were divided into two groups as responders and nonresponders according to the Outcome Measures in Rheumatology (OMERACT) Osteoarthritis Research Society International (OARSI) OA responder criteria.

Demographic and Clinical Assessment:

At the beginning of the study, the age, gender, body mass index (BMI), and pain duration of all participants were recorded. All participants underwent physical examination including a patellar tap test, temperature increase, and range of motion.

Evaluation of Pain and Functional Status:

Visual analog scale (0-100 mm) VAS was used to evaluate pain intensity. The health status of patients with knee OA was evaluated by the Turkish version of the WOMAC Index. The Likert- boxes format of WOMAC was preferred.

Radiographic Evaluation:

The knee anteroposterior (AP) radiographs of all participants in the OA group were taken and evaluated by the researcher and an experienced physical medicine and rehabilitation specialist according to the Kellgren-Lawrence (KL) radiographic staging system. Knee radiographs were not taken for the participants in the control group.

Evaluation of Central Sensitization:

Pain pressure threshold (PPT) measurement and Central Sensitization Inventory (CSI) were used to evaluate central sensitization. The PPT measurement was done on the painful knee in the OA group, on the knee with more severe pain if both knees were painful, and on a randomly determined knee in the control group, on the same side tibialis anterior (TA) muscle and the opposite side forearm. Knee measurement was performed over medial joint spacing, TA muscle measurement was performed 5 cm distal to tuberosity tibia, and forearm measurement was performed 5 cm distal to medial epicondyle on the volar side. Since the medial tibiofemoral compartment is affected more frequently in knee OA, medial joint space was preferred for measurements. TA muscle was evaluated to determine the peripheral spread of pain and the forearm to determine the presence of sensitization at a distant point. All points were selected from places that could be marked according to bone markers so that the measurements could be made from the same points in the participants.

A digital pressure algometer (J-Tech Commander Algometer, USA) was used for the measurements. The hard 1 cm² tip of the algometer was placed perpendicular to the skin on the points to be measured, the pressure was gradually increased until the participant started feeling pain, and the value at the time of pain was recorded. Three measurements were made for each region. During the measurements, the probe was slightly displaced to prevent the sensitization of the region and waited 30 seconds in between. The first measurement was evaluated as a trial learning measurement, the last two measurements were averaged and recorded in Newton/cm2 (N/cm2). It was ensured that the participants did not take analgesics in the last 24 hours before the evaluation, and other medical treatments (antidepressant, pregabalin, etc.) if any, were allowed.

Evaluation of Clinical Conditions Associated with OA and CS:

The possible clinical conditions associated with OA and CS such as neuropathic pain, pain catastrophizing, depression, and sleep problems were also evaluated. The presence of neuropathic pain was assessed by the painDETECT (PD-Q) neuropathic pain questionnaire, pain catastrophizing was assessed by the Pain catastrophizing Scale (PCS), depression was assessed by the Beck Depression Inventory (BDI), and sleep problems were assessed by the Insomnia Severity Index (ISI).

Evaluation of Hyperalgesia:

To investigate the presence of CS in OA patients individually and to show how many of the patients had pressure hyperalgesia, the PPT values from 3 regions of patients were compared separately with the normal reference PPT values obtained from the data of the healthy control group. Reference data were normalized to the specific group means and variances by calculating z-scores recommended by the German Research Network on Neuropathic Pain (DFNS).

Z score = [Value (subject) - Mean (controls)] / Standard deviation (controls)

After the Z transformation, normal distribution of PPT values was achieved. A Z score of 0±1.96 represents 95% of the distribution of the healthy control group's outcomes. Those who were outside the 95% confidence interval of the healthy control group outcomes, i.e. those with a z score of <-1.96 or >1.96, were identified as abnormal. Negative values represent hyperalgesia, positive values represent hypoalgesia.

The Student's t and Mann-Whitney U tests were used to compare variables between the responders and non-responders. Categorical variables were analysed using chi-square test or Fisher's exact chi-square test. Spearman Correlation test was used to investigate the relationship between continuous variables. Logistic regression model was used to evaluate the relationship between groups that responded to and did not respond to treatment and central sensitization. When p<0.05, the results were considered statistically significant.

Sample size determination:

The required sample size was determined by a power analysis before the study. When the investigators accepted the effect size as 0.3145 and the margin of error as 5%, it was concluded that 80 OA patients should be included to reach a power of 80% with 1 degree of freedom chi-square test.

ELIGIBILITY:
Inclusion criteria:

Patient group:

* diagnosed as primary knee osteoarthritis according to the ACR criteria
* between 45-75 years of age
* pain duration of more than 3 months
* pain intensity being 5 or more according to the visual analogue scale (VAS)
* agreeing to participate in the study.

Control group:

* healthy subjects
* between the ages of 45 and 75
* not having pain in the knee and forearm
* not having mechanical, inflammatory, endocrine, degenerative, and systemic co-morbidities that could affect the joints
* agreeing to participate in the study

Exclusion Criteria:

Patient group:

* patients with cervical or lumbar radiculopathy, systemic inflammatory disease, diabetic neuropathy, sensory loss due to chemotherapy or radiotherapy, fibromyalgia or chronic fatigue syndrome
* patients with cognitive impairment or psychiatric illness that prevents cooperation during the evaluation
* patients with a history of previous physical therapy or injections to the knee joints within the last 3 months

Control group:

* subjects with an uncontrolled systemic disease
* subjects with cognitive impairment that prevents cooperation
* subjects with a diagnosis of knee osteoarthritis, chronic painful disease, peripheral neuropathy and rheumatological disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic (Department of Physical Medicine and Rehabilitation, Ankara University, Faculty of Medicine)
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 3 weeks
  Assessment of pain
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Scale | 3 weeks
  Assessment of pain, stiffness, and physical function

SECONDARY OUTCOMES:
Central Sensitization Inventory (CSI) | Baseline
  Assessment of central sensitization
Beck Depression Inventory (BDI) | Baseline
  Assessment of depression
Insomnia Severity Index (ISI) | Baseline
  Assessment of sleep disturbances
Pain Catastrophization Scale (PCS) | Baseline
  Assessment of neuropathic pain
PainDETECT Questionnaire (PD-Q) | Baseline
  Assessment of neuropathic pain
Pressure pain thresholds (PPT) | Baseline
  Assessment of central sensitization

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Gök, Professor, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Cebeci Hospital, Neurorehabilitation Clinic, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Kim MS, Koh IJ, Sohn S, Kang BM, Kwak DH, In Y. Central Sensitization Is a Risk Factor for Persistent Postoperative Pain and Dissatisfaction in Patients Undergoing Revision Total Knee Arthroplasty. J Arthroplasty. 2019 Aug;34(8):1740-1748. doi: 10.1016/j.arth.2019.03.042. Epub 2019 Mar 28. PMID 30992238
- [Result] O'Leary H, Smart KM, Moloney NA, Blake C, Doody CM. Pain sensitization associated with nonresponse after physiotherapy in people with knee osteoarthritis. Pain. 2018 Sep;159(9):1877-1886. doi: 10.1097/j.pain.0000000000001288. PMID 29794610
- [Result] Kim SH, Yoon KB, Yoon DM, Yoo JH, Ahn KR. Influence of Centrally Mediated Symptoms on Postoperative Pain in Osteoarthritis Patients Undergoing Total Knee Arthroplasty: A Prospective Observational Evaluation. Pain Pract. 2015 Jul;15(6):E46-53. doi: 10.1111/papr.12311. Epub 2015 May 16. PMID 25980527
- [Result] Wylde V, Palmer S, Learmonth ID, Dieppe P. The association between pre-operative pain sensitisation and chronic pain after knee replacement: an exploratory study. Osteoarthritis Cartilage. 2013 Sep;21(9):1253-6. doi: 10.1016/j.joca.2013.05.008. PMID 23973138
- [Result] Gervais-Hupe J, Pollice J, Sadi J, Carlesso LC. Validity of the central sensitization inventory with measures of sensitization in people with knee osteoarthritis. Clin Rheumatol. 2018 Nov;37(11):3125-3132. doi: 10.1007/s10067-018-4279-8. Epub 2018 Sep 3. PMID 30178171
- [Result] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Result] Neogi T, Frey-Law L, Scholz J, Niu J, Arendt-Nielsen L, Woolf C, Nevitt M, Bradley L, Felson DT; Multicenter Osteoarthritis (MOST) Study. Sensitivity and sensitisation in relation to pain severity in knee osteoarthritis: trait or state? Ann Rheum Dis. 2015 Apr;74(4):682-8. doi: 10.1136/annrheumdis-2013-204191. Epub 2013 Dec 18. PMID 24351516
- [Result] Uckun AC, Donmez BK, Yurdakul FG, Garip Y, Bodur H. The Role of Pain Catastrophizing and Depression in the Outcomes of Physical Therapy in a Prospective Osteoarthritis Cohort. Pain Physician. 2020 Mar;23(2):209-218. PMID 32214303
- [Result] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Result] Wideman TH, Finan PH, Edwards RR, Quartana PJ, Buenaver LF, Haythornthwaite JA, Smith MT. Increased sensitivity to physical activity among individuals with knee osteoarthritis: relation to pain outcomes, psychological factors, and responses to quantitative sensory testing. Pain. 2014 Apr;155(4):703-711. doi: 10.1016/j.pain.2013.12.028. Epub 2013 Dec 28. PMID 24378879
- [Result] Hochman JR, Davis AM, Elkayam J, Gagliese L, Hawker GA. Neuropathic pain symptoms on the modified painDETECT correlate with signs of central sensitization in knee osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1236-42. doi: 10.1016/j.joca.2013.06.023. PMID 23973136
- [Result] Kurien T, Arendt-Nielsen L, Petersen KK, Graven-Nielsen T, Scammell BE. Preoperative Neuropathic Pain-like Symptoms and Central Pain Mechanisms in Knee Osteoarthritis Predicts Poor Outcome 6 Months After Total Knee Replacement Surgery. J Pain. 2018 Nov;19(11):1329-1341. doi: 10.1016/j.jpain.2018.05.011. Epub 2018 Jun 18. PMID 29920331
- [Result] Tanaka R, Hirohama K. Association of Pain Quality with Pain Catastrophizing and Self-efficacy in People with Knee Osteoarthritis. Prog Rehabil Med. 2018 Feb 7;3:20180002. doi: 10.2490/prm.20180002. eCollection 2018. PMID 32789227
- [Result] Lluch E, Nijs J, Courtney CA, Rebbeck T, Wylde V, Baert I, Wideman TH, Howells N, Skou ST. Clinical descriptors for the recognition of central sensitization pain in patients with knee osteoarthritis. Disabil Rehabil. 2018 Nov;40(23):2836-2845. doi: 10.1080/09638288.2017.1358770. Epub 2017 Aug 2. PMID 28768437
- [Result] Lluch Girbes E, Nijs J, Torres-Cueco R, Lopez Cubas C. Pain treatment for patients with osteoarthritis and central sensitization. Phys Ther. 2013 Jun;93(6):842-51. doi: 10.2522/ptj.20120253. Epub 2013 Feb 7. PMID 23392185